CLINICAL TRIAL: NCT07178405
Title: Effects of Meal Characteristics on Appetite: a Randomized Controlled Trial
Brief Title: Effects of Meal Characteristics on Appetite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 2025-02415-01
Record Dates: First submitted 2025-08-26; First posted 2025-09-17 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Obesity and Obesity-related Medical Conditions; Appetite
Keywords: Appetite; Diet; Intervention; Single meal study
MeSH Terms: conditions — Obesity | interventions — Food, Processed

STUDY DESIGN:
Intervention Model Description: 2*2 factorial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- LL (Experimental): Meal low in energy density, low in ultra-processed food
  Interventions: Other: Meal low in energy density, low in ultra-processed food
- LH (Experimental): Meal low in energy density, high in ultra-processed food
  Interventions: Other: Meal low in energy density, high in ultra-processed food
- HL (Experimental): Meal high in energy density, low in ultra-processed food
  Interventions: Other: Meal high in energy density, low in ultra-processed food
- HH (Experimental): Meal high in energy density, high in ultra-processed food
  Interventions: Other: Meal high in energy density, high in ultra-processed food

INTERVENTIONS:
Other: Meal low in energy density, low in ultra-processed food — Meal low in energy density, low in ultra-processed food
  Other Names: LL
  Arms: LL
Other: Meal low in energy density, high in ultra-processed food — Meal low in energy density, high in ultra-processed food
  Other Names: LH
  Arms: LH
Other: Meal high in energy density, low in ultra-processed food — Meal high in energy density, low in ultra-processed food
  Other Names: HL
  Arms: HL
Other: Meal high in energy density, high in ultra-processed food — Meal high in energy density, high in ultra-processed food
  Other Names: HH
  Arms: HH

SUMMARY:
The overall aim of the study is to determine effects of different meal characteristics on energy intake, eating rate and appetite.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-64 years
* Body mass index (BMI) 18.5-35.0 kg/m2
* Weight stability the last 3 months +/-5%

Exclusion Criteria:

* Food allergies, intolerances or preferences preventing consumption of any products included in the study.
* Unable to sufficiently understand written and spoken Swedish or English to provide written consent and understand information and instructions from the study personal.
* Pregnant, lactating or planning a pregnancy during the study period.
* History of stomach or gastrointestinal conditions or major gastrointestinal surgery (Inflammatory bowel disease, Crohn's disease, malabsorption, colostomy, bowel resection, gastric bypass surgery etc.)
* Type 1 diabetes or type 2 diabetes.
* Drug treated thyroid disorder

  •- Following any weight reduction program or having followed one during the last 6 months prior to screening.
* Medication for weight reduction purpose effecting appetite or fat absorption (e.g. GLP-1 analogues, orlistat)
* Severe dysfunctional eating behavior based on Three Factor Eating Questionnaire

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2025-09-29 (Actual); Primary Completion 2025-11-27 (Actual); Study Completion 2025-11-27 (Actual)

PRIMARY OUTCOMES:
Energy intake | Baseline until 1 hour, or completion of the meal (which ever comes first)
  Energy intake estimated by nutrient calculation of leftover food
Eating rate | Baseline until 1 hour, or completion of the meal (which ever comes first)
  Time it takes to eat the study meal until satisfied

SECONDARY OUTCOMES:
Self-reported appetite | Before, and after the meal (before meal and after 30 minutes, 1hour, 1.5 hours, 2 hours and 4 hours)
  Self-reported appetite, using Visual Analogue Scales
Self-reported prospective energy intake | From 30 min until midnight or bedtime (which ever comes first)
  Self-reported prospective energy intake during the remainder of the day

CONTACTS AND LOCATIONS:
Overall Officials: Linnea Bärebring, PhD, Associate professor, Principal Investigator — Göteborg University
Locations (1):
- University of Gothenburg, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Ethical approvals and legal issues must be considered and resolved before data of individuals can be shared.